CLINICAL TRIAL: NCT04538053
Title: BonE and Joint Infections - Simplifying Treatment in Children Trial
Acronym: BEST
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019.287
Record Dates: First submitted 2020-07-14; First posted 2020-09-03 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Bone Infection; Septic Arthritis; Bone and Joint Infection; Osteomyelitis
MeSH Terms: conditions — Arthritis, Infectious; Osteomyelitis | interventions — Cefazolin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): Children will receive high-dose oral cefalexin 37.5 mg/kg/dose (max 1.5 g) QID 1 to 7 days followed by oral cefalexin 45 mg/kg/dose (max 1.5 g) TDS for a total course of 3 weeks
  Interventions: Drug: Oral cefalexin only
- Standard Therapy (Active Comparator): Children will receive IV cefazolin 50 mg/kg/dose (max 2 g) three-times daily (TDS) or IV flucloxacillin 50 mg/kg/dise (max 2 g) four-times daily (QID) for 1 to 7 days followed by oral cefalexin 45 mg/kg/dose (max 1.5 g) three-times daily (TDS) for a total course of 3 weeks
  Interventions: Drug: IV cefazolin or IV flucloxacillin followed by oral cefalexin

INTERVENTIONS:
Drug: Oral cefalexin only — High-dose oral cefalexin
  Arms: Intervention
Drug: IV cefazolin or IV flucloxacillin followed by oral cefalexin — Standard therapy of IV cefazolin or IV flucloxacillin followed by high dose oral cefalexin
  Arms: Standard Therapy

SUMMARY:
This is a multi- centre trial of children with bone and joint infections (BJIs) at eight major paediatric hospitals in Australia and New Zealand. The primary objective is to establish if in children with acute, uncomplicated BJIs, entirely oral antibiotic treatment is not inferior to initial intravenous (IV) treatment for 1 to 7 days followed by an oral antibiotic course in achieving full recovery 3 months after presentation. Children will be randomly allocated to the 'entirely oral antibiotic' group or the 'standard treatment' group.

DETAILED DESCRIPTION:
Children with acute onset BJIs who present to the participating sites will be enrolled into the trial if eligible (see eligibility criteria) and randomly allocated into two groups. Children in the 'standard treatment group' will receive standard treatment for BJIs, which consists of IV antibiotics for 1-7 days followed by 3 weeks of oral antibiotics. Children in the 'entirely oral treatment group' will receive high dose oral antibiotics, followed by the standard dose of oral antibiotics for 3 weeks. The outcomes of children in each of the two groups will be compared to determine whether BJIs can be treated without needing a course of IV antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 to 18 years with acute, uncomplicated, community-acquired bone and joint infection who fulfil pre-defined clinical criteria.

Exclusion Criteria:

1. Infection due to bacteria resistant to cefalexin or atypical infection (e.g. mycobacterial, fungal)
2. Features of sepsis as defined by the presence of organ dysfunction (defined using definitions within the Pediatric Logistic Organ Dysfunction-2 (PELOD-2) score)
3. Concomitant severe, invasive infection e.g. necrosing fasciitis
4. Complicated infection (e.g. presence of prosthetic material; large subperiosteal (>3mm) or soft tissue abscess without surgical intervention; infection secondary to or complicated by trauma)
5. History of allergy to cephalosporin antibiotics or immediate, severe reaction to penicillins
6. Received more than three IV or oral dose of an antibiotic with activity against the likely bacteria causing the current infection
7. Prior episode of OM or SA
8. Prior condition predisposing to poor absorption (e.g. inflammatory bowel disease, current gastrointestinal symptoms) or complicated disease (e.g. immunodeficiency)
9. Prior enrolment in the trial
10. Current recipient of another investigational product as part of a clinical trial

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 285 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of children assessed as having made a full recovery 3 months | 3 months
  Full recovery is defined by the absence of:
  (i) Clinical features of osteomyelitis or septic arthritis (ii) No episodes of disease recurrence requiring further antibiotic administration after initial treatment.
  Assessment made by a qualified paediatrician.

SECONDARY OUTCOMES:
Proportion of children with with recurrent disease at 6 months. | 6 months
  Proportion of children with recurrence of symptoms and signs after initial recovery requiring further antibiotic administration assessed at 3 months by an independent committee.
Proportion of children with with recurrent disease at 12 months. | 12 months
  Proportion of children with recurrence of symptoms and signs after initial recovery requiring further antibiotic administration assessed at 12 months by an independent committee.
Proportion of children with complications of their disease at 3 months. | 3 months
  Complications assessed by an independent committee defined as:
  (i) residual dysfunction (ii) pain
Proportion of children with complications of their disease at 12 months. | 12 months
  Complications assessed by an independent committee defined as:
  (i) residual poor function (ii) bone death (osteonecrosis) (iii) pain (iv) growth arrest (v) limb deformity
Proportion of children with treatment-related adverse effects (AEs). | Between Day 1-7
  Adverse effects assessed between days 1-7 including:
  (i) Complications of IV access (eg need for replacement, infection, extravasation, drug side effects); or (ii) high-dose oral antibiotics (eg. drug side effects, inability to tolerate the full dose) It will be assessed between day 1-7 (can be at any time during the admission while intravenous antibiotics are prescribed)
Quality of life - Pediatric Quality of Life Inventory (PedsQL) 3 months | 3 months
  PedsQL is an acronym for the Pediatric Quality of Life Inventory. This inventory includes 23 items each scored 0 to 5 . The minimum score is 0 and the maximum score is 92. Lower scores indicate better quality of life. Outcome measures will be reported as median (range).
Quality of life - Child Health Utility Scale (CHU9D) Day 8-14 | Once between Day 8 to Day 14
  CHU9D is an acronym for the Child Health Utility scale. It includes 9 domains scored 0 to 5. The minimum score is 0 and the maximum is 5. The minimum score is 0 and the maximum is 45. Lower scores indicate better quality of life. Outcome measures will be reported as median (range). It will be administered once, and completed any day between Day 8 to Day 14.
Quality of life - Child Health Utility Scale (CHU9D) 12 months | 12 months
  CHU9D is an acronym for the Child Health Utility scale. It includes 9 domains scored 0 to 5. The minimum score is 0 and the maximum is 5. The minimum score is 0 and the maximum is 45. Lower scores indicate better quality of life. Outcome measures will be reported as median (range)
Quality of life - EQ-5d Day 8-14 | Once between Day 8 to Day 14
  EQ-5D is an acronym for the European Quality of Life Five Dimension, it is an instrument which evaluates the generic quality of life. It is a descriptive system with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Outcome measures will be reported as median (range). It will be administered once, and completed any day between Day 8 to Day 14.
Cost effectiveness - cost-effectiveness ratio of all resources at 12 months | 12 months
  The incremental cost-effectiveness ratio will be determined for both arms of the trial. This is a summary measure representing the economic value of the intervention (oral cefalexin), compared with the alternative (IV cefazolin followed by oral cefalexin). Estimated total sum of all hospital and patient/family resources required per patient per treatment course (AUD) collected by the study team at each study visit using a standard questionnaire (e.g. clinical services, medication, hospital and family accommodation, travelling, loss of income, care arrangements for family members). The mean total cost per treatment cost (AUD) will be reported for each arm of the trial.
Treatment adherence - medication reconciliation at 3 weeks | Week 3
  Mean percentage of cefalexin doses taken determined by medication reconciliation (ie. return of any remaining cefalexin) at end of treatment (3 weeks) assessed by the study team/trial pharmacist
Treatment adherence - Medication Adherence Response Scale at 3 weeks | Week 3
  Outcome will be reported as median adherence score (range 5-25).

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Gwee, PhD, Principal Investigator — Murdoch Childrens Research Institute
Locations (10):
- Australia (9):
  - Nepean Hospital, Kingswood, New South Wales
  - John Hunter Children's Hospital, New Lambton Heights, New South Wales
  - Sydney Children's Hospital Network, Sydney, New South Wales
  - The Children's Hospital at Westmead, Sydney, New South Wales
  - Royal Darwin Hospital, Darwin, Northern Territory
  - Queensland Children's Hospital, Brisbane, Queensland
  - Women's and Children's Hospital, Adelaide, South Australia
  - The Royal Children's Hospital, Melbourne, Victoria
  - Perth Children's Hospital, Perth, Western Australia
- Christchurch Hospital, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data set collected for this analysis of the BEST trial will be available six months after publication of the primary outcome.
  The study protocol, analysis plan and consent forms will also be available. The data may be obtained from the Murdoch Children's Research Institute by emailing amanda.gwee@rch.org.au
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Time Frame: 6 months after publication of primary outcome
Access Criteria: Prior to releasing any data the following are required: a data access agreement must be signed between relevant parties, the BEST Trial Principle and Associate Investigators must see and approve the analysis plan describing how the data will be analysed, there must be an agreement around appropriate acknowledgement and any additional costs involved must be covered. Data will only be shared with a recognised research institution which has approved the proposed analysis plan.
URL: https://www.mcri.edu.au/research/core-facilities-services/melbourne-children-trials-centre